CLINICAL TRIAL: NCT02551055
Title: An Umbrella Study to Evaluate MLN1117 in Combination With Taxanes (Docetaxel or Paclitaxel) and Other Investigational Anticancer Agents for the Treatment of Patients With Previously Treated Advanced and Metastatic Gastric and Gastroesophageal Adenocarcinoma
Brief Title: MLN1117 in Combination With Docetaxel, Paclitaxel, and Other Investigational Anticancer Agents to Treat Participants With Gastric and Gastroesophageal Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision; No Safety Or Efficacy Concerns.
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C032-6001 (MLN1117-1003); 2015-001032-38 (EudraCT Number); U1111-1166-8653 (Registry Identifier: WHO); REec-2016-2039 (Other: REEC)
Record Dates: First submitted 2015-09-02; First posted 2015-09-16 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Advanced and Metastatic Gastric or Gastroesophageal Adenocarcinoma
Keywords: Drug Therapy
MeSH Terms: interventions — serabelisib; TAK-659; MLN 8237; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- MLN1117 300 mg + Alisertib (Experimental): MLN1117 300 mg, tablets, orally, once daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15, 16, 17; 22, 23, and 24) and 4 days off per week and alisertib 40 mg, tablets, orally, twice daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15,16, and 17) and 4 days off per week on Weeks 1-3, and 1 week off in 28-day treatment cycles until PD or unacceptable toxicity.
  Interventions: Drug: MLN1117; Drug: Alisertib
- MLN1117 600 mg + Alisertib (Experimental): MLN1117 600 mg, tablets, orally, once daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15, 16, 17; 22, 23, and 24) and 4 days off per week and alisertib 40 mg, tablets, orally, twice daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15,16, and 17) and 4 days off per week on Weeks 1-3, and 1 week off in 28-day treatment cycles until PD or unacceptable toxicity.
  Interventions: Drug: MLN1117; Drug: Alisertib
- MLN1117 300 mg + Paclitaxel (Experimental): MLN1117 300 mg, tablets, orally, once daily for 3 days on (Days 2, 3, 4; 9, 10, 11; 16, 17, 18; 23, 24, and 25) and 4 days off per week and paclitaxel 80 mg/m^2, infusion, intravenously, once weekly on (Days 1, 8, and 15) and 1 week off, in 28-day treatment cycles until PD or unacceptable toxicity.
  Interventions: Drug: MLN1117; Drug: Paclitaxel
- MLN1117 600 mg + Paclitaxel (Experimental): MLN1117 600 mg, tablets, orally, once daily for 3 days on (Days 2, 3, 4; 9, 10, 11; 16, 17, 18; 23, 24, and 25) and 4 days off per week and paclitaxel 80 mg/m^2, infusion, intravenously, once weekly on (Days 1, 8, and 15) and 1 week off, in 28-day treatment cycles until PD or unacceptable toxicity.
  Interventions: Drug: MLN1117; Drug: Paclitaxel
- MLN1117 300 mg + TAK-659 (Experimental): MLN1117 300 mg, tablets, orally, once daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15, 16, 17; and 22, 23, and 24) and 4 days off per week and TAK-659 100 mg (as determined in study C34001 [NCT02000934]), tablets, orally, once daily, in 28-day treatment cycles until progressive disease (PD) or unacceptable toxicity.
  Interventions: Drug: MLN1117; Drug: TAK-659; Drug: Docetaxel
- MLN1117 200 mg + Docetaxel (Experimental): MLN1117 200 mg, orally, once daily for 3 days on (Days 2, 3, 4; 9, 10, 11; 16, 17, and 18) and 4 days off per week and docetaxel 75 mg/m^2, infusion, intravenously, on Day 1 once every 3 weeks in 21-day treatment cycles until PD or unacceptable toxicity.
  Interventions: Drug: MLN1117; Drug: Docetaxel
- MLN1117 300 mg + Docetaxel (Experimental): MLN1117 300 mg, orally, once daily for 3 days on (Days 2, 3, 4; 9, 10, 11; 16, 17, and 18) and 4 days off per week and docetaxel 75 mg/m^2, infusion, intravenously, on Day 1 once every 3 weeks in 21-day treatment cycles until PD or unacceptable toxicity.
  Interventions: Drug: MLN1117

INTERVENTIONS:
Drug: MLN1117 — MLN1117 Tablets
  Other Names: TAK-117
Drug: TAK-659 — TAK-659 Tablets
  Arms: MLN1117 300 mg + TAK-659
Drug: Alisertib — Alisertib Tablets
  Other Names: MLN8237
  Arms: MLN1117 300 mg + Alisertib; MLN1117 600 mg + Alisertib
Drug: Paclitaxel — Paclitaxel intravenous infusion
  Arms: MLN1117 300 mg + Paclitaxel; MLN1117 600 mg + Paclitaxel
Drug: Docetaxel — Docetaxel intravenous infusion
  Arms: MLN1117 200 mg + Docetaxel; MLN1117 300 mg + TAK-659

SUMMARY:
The purpose of this study is to evaluate the maximum tolerated dose (MTD) or recommended Part 2 dose, safety and efficacy of MLN1117 (TAK-117) in combination with docetaxel, paclitaxel, investigational TAK-659 or investigational alisertib in adult participants with advanced and metastatic gastric or gastroesophageal adenocarcinoma. The study consists of a dose escalation phase (Part 1) and a dose expansion phase (Part 2).

DETAILED DESCRIPTION:
The drug being tested in this study is called MLN1117. MLN1117 is being tested to treat people who have locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma. This study will look at the dose-limiting toxicity and response to treatment in participants who take MLN1117 in combination with TAK-659, alisertib, paclitaxel, or docetaxel.

The study will enroll 32 participants in the dose escalation phase (Part 1) and 118 participants in the dose expansion phase (Part 2). Participants will be assigned to 1 of the 7 treatment groups:

* MLN1117 300 mg+Alisertib
* MLN1117 600 mg+Alisertib
* MLN1117 300 mg+Paclitaxel
* MLN1117 600 mg+Paclitaxel
* MLN1117 300 mg+TAK-659
* MLN1117 200 mg+Docetaxel
* MLN1117 300 mg+Docetaxel

In Part 1, the dose of MLN1117 will be increased step by step. All participants will be asked to take tablets of MLN1117 for 3 days on and 4 days off per week in 28-day treatment cycles or 21-day treatment cycles when given in combination with the other companion drugs.

This multi-center trial will be conducted in Spain and United States. The overall time to participate in this study is 10 months for Part 1 and 24 months for Part 2. Participants will make multiple visits to the clinic, and be contacted by telephone, e-mail or mail every 12 weeks for up to 6 months or 1 year after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Part 1 and Part 2

1. Is male or female aged 18 years or older at the time of consent.
2. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 14 days before enrollment.
3. Has adequate organ and hematologic function as evidenced by the following laboratory values within 14 days before enrollment:

   * Absolute neutrophil count (ANC) ≥1.5x10^9/L.
   * Platelet count ≥100x10^9/L.
   * Hemoglobin ≥9 g/dL (Transfusions are allowed to reach this hemoglobin level).
   * Serum creatinine ≤1.5 times the upper limit of the normal range (ULN) or creatinine clearance ≥50 mL/min either as estimated by the Cockcroft-Gault equation or based on urine collection (12 or 24 hours).
   * Total bilirubin ≤1.5×ULN.
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5×ULN.
4. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception at the same time, from the time of signing the informed consent form through 30 days after the last dose of study drug (with the exception of those participants assigned to TAK-659, for whom the duration required is 180 days), or for as long as mandated by local labeling for docetaxel and paclitaxel, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant, from the time of signing the informed consent form through 30 days after the last dose of study drug (with the exception of those participants assigned to TAK-659, for whom the duration required is 180 days), or for as long as mandated by local labeling for docetaxel and paclitaxel. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

   Male participants, even if surgically sterilized (ie, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug (with the exception of those participants assigned to TAK-659, for whom the duration required is 180 days), or for as long as mandated by local labeling for docetaxel and paclitaxel, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant during the entire study treatment period and through 120 days after the last dose of study drug (with the exception of those participants assigned to TAK-659, for whom the duration required is 180 days) or for as long as mandated by local labeling for docetaxel and paclitaxel. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
5. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
6. Has suitable venous access for the study-required blood sampling (ie, pharmacokinetic (PK) sampling, circulating tumor deoxyribonucleic acid [DNA]).

Part 1 only

1. Has a histologically confirmed diagnosis of advanced solid tumor, including but not limited to gastric or gastroesophageal junction adenocarcinoma.
2. Has radiographically or clinically evaluable disease. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 is not required.
3. Is relapsed or refractory with no effective therapeutic options available.

Part 2 only

1. Has a histologically confirmed diagnosis of metastatic or locally advanced adenocarcinoma of the stomach or gastroesophageal junction (Stage IIIb or IV according to International Union Against Cancer [UICC] tumor, node, metastases [TNM] classification, 7th edition).
2. Has at least 1 measurable tumor lesion per RECIST Version 1.1 by radiographic techniques (computed tomography [CT] or magnetic resonance imaging [MRI]).
3. Has receipt of 1 prior systemic chemotherapy regimen for advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction with documented progressive disease (PD).
4. Has archived or fresh tumor biopsy samples obtained during screening sufficient for Epstein-Barr virus (EBV) testing and genotyping.

Exclusion Criteria:

Part 1 and Part 2

1. Has received prior systemic anticancer therapies or other investigational agents within 2 weeks before the first administration of study drug or has failed to recover from the adverse drug effects of prior therapies (to ≤Grade 1 or to a level meeting inclusion criteria). For prior therapies with a half-life longer than 3 days, the interval must equal minimally 28 days before the first administration of study drug and the participant must have documented PD.
2. Has radiotherapy within 14 days before enrollment.
3. Has fasting glucose ≥130 mg/dL. Poorly controlled diabetes mellitus (glycosylated hemoglobin [HbA1c] >7.0%). Participants with a history of transient glucose intolerance due to corticosteroid administration are allowed.
4. Has received strong cytochrome P-450 (CYP) 3A4 inducers/inhibitors within 7 days before the first administration of study drug or has conditions that require the concomitant use of CYP3A4 inducers/inhibitors during the course of the study.
5. For TAK-659 (Cohort A) only: Is receiving treatment with medications that are known to be inhibitors or inducers of P-glycoprotein (P-gp). Baseline lipase >ULN. Participants not fulfilling these exclusion criteria can be enrolled in other cohorts (Part 1 only).
6. Has taken proton pump inhibitors within 7 days before the first administration of study drug or has conditions that require the concomitant use of proton pump inhibitors during the course of the study.
7. Has signs of peripheral neuropathy ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade 2.
8. Has symptomatic brain metastases or brain metastases with a stable neurologic status for <2 weeks after completion of the definitive therapy and steroids.
9. Has systemic infection requiring intravenous (IV) antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
10. Has known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection. Testing for these agents is not required in the absence of clinical findings or suspicion.
11. Has known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerability of orally administered study drug, including difficulty swallowing tablets; diarrhea >Grade 1 despite supportive therapy; or prior total gastrectomy.
12. Has clinically significant comorbidities, such as uncontrolled pulmonary disease, known impaired cardiac function or clinically significant cardiac disease, active central nervous system disease, or any other condition that could compromise the participant's participation in the study.

    • Known impaired cardiac function or clinically significant cardiac disease includes: evidence of currently uncontrolled cardiovascular conditions (including arrhythmias, angina, pulmonary hypertension, acute ischemia or active conduction system abnormalities); current history of New York Heart Association Class III or IV heart failure; acute myocardial infarction within 6 months before starting study drug; baseline QT interval corrected for heart rate (QTc) ≥Grade 1 according to NCI CTCAE Version 4.03 criteria; or abnormalities on baseline 12-lead ECG that are considered clinically significant per the investigator.
13. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before the first dose of study drug.
14. Participants with bilirubin >ULN, or AST and/or ALT >1.5 X ULN concomitant with alkaline phosphatase >2.5 X ULN cannot be allocated to Cohort D (MLN1117+docetaxel) in Part 1 and are not eligible for Part 2 if they are also EBV negative.

Part 2 only

1. Has prior treatment with any of the following:

* An Aurora A-targeted agent (not eligible for randomization in Cohorts B, C, or D, but eligible for Cohort A if EBV positive).
* A docetaxel- or paclitaxel-containing chemotherapy regimen (not eligible for randomization in Cohorts B, C, or D, but eligible for Cohort A if EBV positive).
* A spleen tyrosine kinase (SYK) inhibitor (MLN1117+TAK-659 arm only).
* A phosphoinositide 3-kinase (PI3K) or serine/threonine kinase, also known as protein kinase B or PKB (AKT) inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (6):
- United States (5):
  - Lake Success, New York
  - New York, New York
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
- Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in Spain and the United States from 15 October 2015 to 18 January 2017.
Pre-assignment Details: Participants with solid advanced tumors were enrolled in Part 1 to receive MLN1117 along with alisertib, paclitaxel, TAK-659 and docetaxel in 1 of 7 treatment regimens. In Part 2, participants with gastric or gastroesophageal junction adenocarcinoma were to be enrolled, however, study terminated before initiation of part 2.
Groups:
- MLN1117 300 mg + Alisertib: MLN1117 300 mg, tablets, orally, once daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15, 16, 17; 22, 23, and 24) and 4 days off per week and alisertib 40 mg, tablets, orally, twice daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15,16, and 17) and 4 days off per week on Weeks 1-3, and 1 week off in 28-day treatment cycles until PD or unacceptable toxicity (up to 12 cycles).
- MLN1117 600 mg + Alisertib: MLN1117 600 mg, tablets, orally, once daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15, 16, 17; 22, 23, and 24) and 4 days off per week and alisertib 40 mg, tablets, orally, twice daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15,16, and 17) and 4 days off per week on Weeks 1-3, and 1 week off in 28-day treatment cycles until PD or unacceptable toxicity (up to 10 cycles).
- MLN1117 300 mg + Paclitaxel: MLN1117 300 mg, tablets, orally, once daily for 3 days on (Days 2, 3, 4; 9, 10, 11; 16, 17, 18; 23, 24, and 25) and 4 days off per week and paclitaxel 80 mg/m^2, infusion, intravenously, once weekly on (Days 1, 8, and 15) and 1 week off, in 28-day treatment cycles until PD or unacceptable toxicity (up to 6 cycles).
- MLN1117 600 mg + Paclitaxel: MLN1117 600 mg, tablets, orally, once daily for 3 days on (Days 2, 3, 4; 9, 10, 11; 16, 17, 18; 23, 24, and 25) and 4 days off per week and paclitaxel 80 mg/m^2, infusion, intravenously, once weekly on (Days 1, 8, and 15) and 1 week off, in 28-day treatment cycles until PD or unacceptable toxicity (up to 3 cycles).
- MLN1117 300 mg + TAK-659: MLN1117 300 mg, tablets, orally, once daily for 3 days on (Days 1, 2, 3; 8, 9, 10; 15, 16, 17; and 22, 23, and 24) and 4 days off per week and TAK-659 100 mg (as determined in study C34001 [NCT02000934]), tablets, orally, once daily, in 28-day treatment cycles until progressive disease (PD) or unacceptable toxicity (up to 3 cycles).
- MLN1117 200 mg + Docetaxel: MLN1117 200 mg, orally, once daily for 3 days on (Days 2, 3, 4; 9, 10, 11; 16, 17, and 18) and 4 days off per week and docetaxel 75 mg/m^2, infusion, intravenously, on Day 1 once every 3 weeks in 21-day treatment cycles until PD or unacceptable toxicity (up to 1 cycle).
- MLN1117 300 mg + Docetaxel: MLN1117 300 mg, orally, once daily for 3 days on (Days 2, 3, 4; 9, 10, 11; 16, 17, and 18) and 4 days off per week and docetaxel 75 mg/m^2, infusion, intravenously, on Day 1 once every 3 weeks in 21-day treatment cycles until PD or unacceptable toxicity (up to 2 cycles).
- Part 2: Participants entered Part 2 of the study were to be screened to determine EBV-positive or EBV-negative solid tumors. EBV-positive participants were to receive MLN1117+TAK-659 (Cohort A). EBV-negative participants were to be randomized to other treatment cohorts: MLN1117+alisertib (Cohort B), MLN1117+paclitaxel (Cohort C), or MLN1117+docetaxel (Cohort D).
Period: Overall Study
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel | Part 2
Started | 4 | 6 | 3 | 6 | 7 | 2 | 4 | 0
Completed | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Not Completed | 4 | 6 | 2 | 5 | 7 | 1 | 3 | 0
Not completed — Death | 2 | 4 | 2 | 2 | 2 | 1 | 2 | 0
Not completed — Study Terminated by Sponsor | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Reason not specified | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population is defined as all participants who received at least 1 dose of any study drug. Participants are analyzed according to the treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel | Total
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (7.94) | 59.0 (4.86) | 65.3 (13.28) | 62.2 (11.82) | 62.3 (9.16) | 65.5 (4.95) | 62.3 (9.95) | 62.0 (8.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 5 | 7 | 2 | 2 | 25
  Male | 1 | 3 | 0 | 1 | 0 | 0 | 2 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 4 | 6 | 3 | 5 | 6 | 2 | 3 | 29
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 4 | 2 | 6 | 6 | 1 | 4 | 27
  Black or African American | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 4
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 3 | 3 | 6 | 2 | 4 | 27
  Spain | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 5
Height [Mean (Standard Deviation); unit: cm] | 162.90 (14.178) | 165.50 (10.145) | 159.80 (4.513) | 162.83 (15.108) | 158.76 (6.662) | 154.95 (7.142) | 166.25 (16.674) | 162.07 (10.939)
Weight [Mean (Standard Deviation); unit: kg] | 77.75 (15.314) | 71.63 (19.725) | 74.07 (12.756) | 82.38 (25.474) | 65.53 (13.046) | 75.45 (43.911) | 68.28 (21.403) | 73.13 (19.400)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body Surface Area (m^2) = sqrt [height (cm)* weight (kg)/3600]
  m^2 | 1.825 (0.2814) | 1.802 (0.2863) | 1.809 (0.1638) | 1.917 (0.3496) | 1.694 (0.1790) | 1.768 (0.5769) | 1.767 (0.3734) | 1.796 (0.2796)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Cycle 1 Dose Limiting Toxicity (DLT) in Part 1
Description: Toxicity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0. DLT defined as any of following considered related to any of treatment by investigator: Grade 4 neutropenia (absolute neutrophil count <500 cells/mm^3) for >7 days; ≥ Grade 3 neutropenia with coincident fever or infection; Grade 4 thrombocytopenia for >7 days; Grade 3 thrombocytopenia with clinically significant bleeding; Platelet count <10,000/mm^3 at any time; Delay in initiation of subsequent therapy cycle by >7 days due to treatment-related toxicity; ≥Grade 3 nonhematological toxicity except Grade 3 arthralgia/myalgia, fatigue that lasts <1 month, diarrhea, fasting hyperglycemia lasting ≤14 days, rash lasting ≤7 days and any other Grade 3 nonhematological toxicity that could be safely, reliably controlled to ≤Grade 1 with appropriate treatment; ≥ Grade 2 nonhematologic toxicities that are considered by investigator to be related to study drugs and dose-limiting.
Time Frame: Up to Cycle 1 (28 days for MLN1117+TAK-659, MLN1117+Alisertib, MLN1117+Paclitaxel or 21 days for MLN1117+Docetaxel)
Population: DLT-evaluable population defined as all participants in Part 1 of study who either experience DLT during Cycle 1 or complete treatment with at least 75% of the planned doses of MLN1117 and the combination partner, and have sufficient follow-up data for the investigators and sponsor to determine whether DLT occurred.
Measure: Number; unit: participants
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4
participants | 0 | 1 | 0 | 0 | 1 | 0 | 1

2. Primary Outcome: Number of Participants With at Least 1 Treatment-Emergent Adverse Event (TEAE) in Part 1
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately up to 366 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4
participants | 4 | 6 | 3 | 6 | 7 | 2 | 4

3. Primary Outcome: Number of Participants With at Least 1 ≥ Grade 3 TEAE in Part 1
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAE is defined as an adverse event with an onset that occurs after receiving study drug. There are 5 grades of the CTCAE; "grade" refers to severity. Grade 5 is the most severe, grade 1 is the least severe. As per version 4.0 of the CTCAE, Grade 3 = AE with severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4 = AE with life-threatening consequences; urgent intervention indicated and Grade 5 = Death related to AE.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately up to 366 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4
participants | 4 | 4 | 2 | 2 | 6 | 2 | 4

4. Primary Outcome: Number of Participants With at Least 1 Treatment-Emergent Serious Adverse Event (SAE) in Part 1
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; or a medically important event. TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately up to 366 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4
participants | 2 | 3 | 1 | 2 | 5 | 2 | 4

5. Primary Outcome: Number of Participants With at Least 1 Dose Modification Due to AE in Part 1
Description: A decision regarding which study drug requires dose modification is dependent upon the toxicity, its onset, and time course. The causal relationship of each AE should will be assessed in relation to MLN1117 and to the combination agent in each cohort so that dose modifications can be made accordingly. Intrapatient dose reductions of MLN1117 are not permitted during Part 1 Cycle 1 unless the participant experiences a DLT attributed to MLN1117. Per dose modification guidelines, participants who have the study drug held because of treatment related or possibly related AEs may resume study drug treatment after resolution of the AE but may either maintain the same dose level or have doses of study drug reduced (dose reduction) by at least 1 dose level and if needed, by 2 dose levels. When a dose reduction of MLN1117 occurs, the MLN1117 dose will be reduced to the next lower dose that has been established as a safe dose during dose escalation (Part 1).
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately up to 366 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4
participants | 0 | 1 | 1 | 0 | 4 | 0 | 1

6. Primary Outcome: Overall Response Rate in Part 2
Description: Overall response is defined as complete response (CR) plus partial response (PR) according to Response Evaluation Criteria in Solid tumors (RECIST) version 1.1 criteria. According to RECIST: CR is defined as disappearance of all target lesions and PR is defined as 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Days 25-28 for MLN1117+TAK-659, MLN1117+Alisertib, and MLN1117+Paclitaxel and Days 18-21 for MLN1117+Docetaxel of Cycles 2, 4, 6; every other cycle until study discontinuation due to disease progression, unacceptable toxicity, or death (up to 336 days)
Population: Study was terminated before the initiation of Part 2 of the study.
Arm/Group | Part 2
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With at Least 1 TEAE and Serious TEAE in Part 1 and 2
Description: as for outcome 4
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately up to 366 days)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel | Part 2
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4 | 0
participants
  AE | 4 | 6 | 3 | 6 | 7 | 2 | 4 |
  SAE | 2 | 3 | 1 | 2 | 5 | 2 | 4 |

8. Secondary Outcome: Number of Participants With Dose Delays, Dose Reductions, and Dose Interruptions Due To AE in Part 1 and 2
Description: Per dose modification guidelines, participants who have the study drug held because of treatment related or possibly related AEs may resume study drug treatment after resolution of the AE but may either maintain the same dose level or have doses of study drug reduced (dose reduction) by at least 1 dose level and if needed, by 2 dose levels.
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately up to 366 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel | Part 2
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4 | 0
Participants
  Dose delay due to AE | 0 | 0 | 0 | 0 | 1 | 0 | 0 |
  Dose reduction due to AE | 0 | 1 | 1 | 0 | 4 | 0 | 1 |
  Dose interruption due to AE | 0 | 0 | 1 | 0 | 0 | 0 | 0 |

9. Secondary Outcome: Progression-Free Survival (PFS) Based on RECIST Criteria V 1.1 Assessment in Part 2
Description: PFS is defined as the time from the date of randomization to the date of first documentation of Progressive disease (PD) or death due to any cause, whichever occurs first. PD is defined as an increase of >=20% from the nadir (or baseline, if it represents the point at which the sum of target disease was lowest).
Time Frame: as for outcome 6
Population: Study was terminated before the initiation of Part 2 of the study.
Arm/Group | Part 2
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Participants With Disease Control Based on RECIST Criteria V 1.1 Assessment in Part 2
Description: Disease control rate is defined as the percentage of participants with complete response (CR) + Partial response (PR) + stable disease (SD) according to RECIST version 1.1 criteria. CR is defined as disappearance of all target lesions, PR is defined as 30% decrease in the sum of the longest diameter of target lesions and SD is defined as not qualifying for CR, PR, or PD.
Time Frame: as for outcome 6
Population: Study was terminated before the initiation of Part 2 of the study.
Arm/Group | Part 2
Number analyzed (Participants) | 0

11. Secondary Outcome: Duration of Response (DOR) Based on RECIST Criteria V 1.1 Assessment in Part 2
Description: DOR is defined as the time from the date of first documentation of a response to the date of first documentation of PD according to RECIST version 1.1 criteria. PD is defined as 20% increase in the sum of the longest diameter of target lesions for measurable neoplastic disease.
Time Frame: as for outcome 6
Population: Study was terminated before the initiation of Part 2 of the study.
Arm/Group | Part 2
Number analyzed (Participants) | 0

12. Secondary Outcome: Time to Disease Progression (TTP) Based on RECIST Criteria V 1.1 Assessment in Part 2
Description: TTP is defined as the time from the date of randomization to the date of first documentation of PD. PD is defined as 20% increase in the sum of the longest diameter of target lesions for measurable neoplastic disease.
Time Frame: as for outcome 6
Population: Study was terminated before the initiation of Part 2 of the study.
Arm/Group | Part 2
Number analyzed (Participants) | 0

13. Secondary Outcome: Overall Survival (OS) Based on RECIST Criteria V 1.1 Assessment
Description: OS is defined as the time from the date of randomization to the date of death.
Time Frame: From randomization up to end of Part 2, then every 12 weeks until participant death or until 1 year after the last dose of study drug, whichever occurs first (up to 336 days)
Population: Study was terminated before the initiation of Part 2 of the study.
Arm/Group | Part 2
Number analyzed (Participants) | 0

14. Secondary Outcome: Plasma Concentration of MLN1117-1003
Time Frame: MLN1117 300 mg + Alisertib arms: Cycle 1 Day 3; MLN1117 300 mg + Paclitaxel arms and MLN1117 200 mg + Docetaxel arms: Cycle 1 Day 2; MLN1117 300 mg + TAK-659 arm: Cycle 1 Days 1 and 17
Population: Pharmacokinetic (PK) evaluable population included all participants in Part 1 (dose escalation of the study for whom there were sufficient dosing and MLN1117 concentration-time data was available).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel
Number analyzed (Participants) | 4 | 6 | 3 | 6 | 7 | 2 | 4
ng/mL
  Day 1: Predose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 0.00 (0.000) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 1: 0.5 Hour Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 675.04 (816.641) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 1: 1 Hour Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 2171.00 (1840.041) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 1: 2 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 3054.14 (1811.084) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 1: 3 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 3315.29 (1521.130) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 1: 4 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 3164.71 (1522.096) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 1: 6 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 2726.71 (1259.976) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 1: 8 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 2466.29 (1112.350) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 1: 24 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 1045.17 (642.781) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 2: Predose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 0.00 (0.000) | 0.00 (0.000) | NA (NA) — Data was not analyzed at this timepoint. | 0.00 (0.000) | 0.00 (0.000)
  Day 2: 0.5 Hour Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 1762.00 (1295.728) | 1701.17 (1407.015) | NA (NA) — Data was not analyzed at this timepoint. | 3240.00 (1230.366) | 1333.05 (1970.336)
  Day 2: 1 Hour Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 3840.00 (747.195) | 3261.83 (2879.952) | NA (NA) — Data was not analyzed at this timepoint. | 3165.00 (1859.691) | 1554.00 (2042.092)
  Day 2: 2 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 4066.67 (322.542) | 3934.00 (3419.860) | NA (NA) — Data was not analyzed at this timepoint. | 4615.00 (4433.560) | 1456.23 (1577.178)
  Day 2: 3 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 3653.33 (325.628) | 3753.50 (3324.071) | NA (NA) — Data was not analyzed at this timepoint. | 4355.00 (4362.849) | 1598.75 (1269.397)
  Day 2: 4 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 3206.67 (256.970) | 3994.67 (3191.500) | NA (NA) — Data was not analyzed at this timepoint. | 3725.00 (3542.605) | 1475.75 (1062.242)
  Day 2: 6 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 2720.00 (10.000) | 4311.67 (2752.595) | NA (NA) — Data was not analyzed at this timepoint. | 3085.00 (2920.351) | 1417.75 (907.208)
  Day 2: 8 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 2536.67 (87.369) | 3246.00 (2026.285) | NA (NA) — Data was not analyzed at this timepoint. | 3025.00 (2807.214) | 1443.25 (992.241)
  Day 2: 24 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 592.67 (38.527) | 1279.83 (1238.550) | NA (NA) — Data was not analyzed at this timepoint. | 717.00 (668.923) | 420.80 (477.731)
  Day 3: Predose | 2177.50 (1453.717) | 3178.82 (2696.065) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 3: 0.5 Hour Postdose | 3225.00 (693.229) | 4554.80 (3431.547) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 3: 1 Hour Postdose | 5010.00 (1376.590) | 5070.60 (3278.807) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 3: 2 Hours Postdose | 5007.50 (1192.347) | 6235.80 (4139.804) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 3: 3 Hours Postdose | 4815.00 (810.535) | 5650.00 (3995.103) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 3: 4 Hours Postdose | 4797.50 (1240.225) | 4719.20 (3100.983) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 3: 6 Hours Postdose | 4777.50 (1753.024) | 4501.80 (2904.730) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 3: 8 Hours Postdose | 4320.00 (1862.078) | 4354.80 (2836.444) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 3: 24 Hours Postdose | 2217.33 (1604.245) | 2357.42 (1806.031) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 17: Predose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 978.33 (1519.070) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 17: 0.5 Hour Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 2893.67 (1738.859) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 17: 1 Hour Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 5596.67 (387.599) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 17: 2 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 5583.33 (1146.575) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 17: 3 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 5116.67 (1608.426) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 17: 4 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 5066.67 (2009.784) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 17: 6 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 4293.33 (1654.398) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.
  Day 17: 8 Hours Postdose | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint. | 4330.00 (2606.971) | NA (NA) — Data was not analyzed at this timepoint. | NA (NA) — Data was not analyzed at this timepoint.

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug. Related SAEs could be reported at any time after discontinuation.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Laboratory finding that are considered clinically significant, drive dose modifications or the use of concomitant medications, are considered AEs.
Arm/Group | MLN1117 300 mg + Alisertib | MLN1117 600 mg + Alisertib | MLN1117 300 mg + Paclitaxel | MLN1117 600 mg + Paclitaxel | MLN1117 300 mg + TAK-659 | MLN1117 200 mg + Docetaxel | MLN1117 300 mg + Docetaxel
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 1/3 | 1/6 | 1/7 | 1/2 | 2/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/6 | 1/3 | 2/6 | 5/7 | 2/2 | 4/4
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 3/3 | 6/6 | 7/7 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN1117 300 mg + Alisertib (N=4) | MLN1117 600 mg + Alisertib (N=6) | MLN1117 300 mg + Paclitaxel (N=3) | MLN1117 600 mg + Paclitaxel (N=6) | MLN1117 300 mg + TAK-659 (N=7) | MLN1117 200 mg + Docetaxel (N=2) | MLN1117 300 mg + Docetaxel (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN1117 600 mg+Paclitaxel and is not related; One treatment-emergent death occurred during treatment with MLN1117 300 mg+TAK-659 and is not related.
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with MLN1117 300 mg+Docetaxel and is not related.
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN1117 300 mg+Paclitaxel and is not related
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with MLN1117 300 mg+Docetaxel and is not related.
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with MLN1117 200 mg+Docetaxel and is not related.
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN1117 300 mg + Alisertib (N=4) | MLN1117 600 mg + Alisertib (N=6) | MLN1117 300 mg + Paclitaxel (N=3) | MLN1117 600 mg + Paclitaxel (N=6) | MLN1117 300 mg + TAK-659 (N=7) | MLN1117 200 mg + Docetaxel (N=2) | MLN1117 300 mg + Docetaxel (N=4)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 4 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 3 | 4 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 4 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 0 | 1 | 2 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 1 | 0 | 1 | 1 | 2
Chills (General disorders) | 0 | 2 | 1 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 1 | 2 | 0 | 1 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychomalacia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 3 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 3 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis in device (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, the pharmacokinetic data collected was not processed further. Therefore, the planned secondary endpoints of PK summary statistics are not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT02551055/Prot_SAP_000.pdf